CLINICAL TRIAL: NCT01073657
Title: Supporting Education Goals of OIF/OEF Veterans With PTSD: Pilot Process & Outcome
Brief Title: Supported Education Pilot
Acronym: SEd
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PPO 09-254
Record Dates: First submitted 2010-02-18; First posted 2010-02-23 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-09

CONDITIONS: PTSD
Keywords: Rehabilitation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supported Education (Experimental): Veterans received supported education services. A Veteran peer met weekly as needed with a subject for up to six months in a psycho-social rehabilitation service for meeting education goals. Goals included choosing a college, getting admitted or enrolled, and maintaining enrollment and completing classes.
  Interventions: Other: Supported Education
- General Peer Support (Active Comparator): Matched attention was provided by a Veteran peer who met weekly with Veterans but who focused on help with any personal goal (eg, employment, housing) but not on education.
  Interventions: Other: General Peer Support

INTERVENTIONS:
Other: Supported Education — Rehabilitation counseling using peers to achieve educational goals
  Other Names: Psychosocial Rehabilitation
  Arms: Supported Education
Other: General Peer Support — Matched peer support for any personal goal other than education
  Arms: General Peer Support

SUMMARY:
The goal of this project is to gather data necessary for a full scale trial of a supported education service for OIF/OEF veterans with PTSD. Forty Veterans with PTSD will be randomly assigned to an intervention group (N=20) that receives a weekly supported education intervention and a control group that receives services as usual plus an hour of attentive intervention not focused on education. We will assess and compare the number of hours of participation in community education settings and on acquiring an educational goal for the Veterans in each group.

DETAILED DESCRIPTION:
Goal: The goal of this project is to gather data on feasibility and effect size necessary for a full scale trial of a supported education service for Operation Iraq and Enduring Freedom (OIF/OEF) veterans with PTSD that will contribute to its evidence-base. Supported education is a rehabilitation and recovery based intervention that is new to VHA services and that responds to an expressed but unmet need among these warriors with war-related trauma. We propose to conduct a pilot of a supported education service and employ a process and outcome evaluation.

Anticipated Impacts on Veterans Healthcare: Veterans with post traumatic stress disorder (PTSD) possess educational aspirations. Due to limited education and disability adjustment, many such veterans unsuccessfully locate employment or obtain entry level jobs with limited advancement opportunities. Even with current GI Bill funding increases, veterans experience non-financial barriers to their pursuit of educational goals. Supported education is a strategy developed within the civilian population that facilitates skill, career, and educational goals within post-secondary educational settings. It has been shown to increase educational engagement, participation, and completion, as well as improve empowerment and school efficacy. We hypothesize that supported education tailored to returning Veterans will result in similar outcomes.

Aims and Objectives: The goal of this project is to gather data necessary for a full scale trial of a supported education service for OIF/OEF veterans with PTSD. The following are the aims and objectives:

Aim 1: Using a randomized controlled design, assess the magnitude of the effect of a supported education service on hours of participation in community educational settings and on acquiring an educational goal. Objective: Assess the number of hours of participation in community education settings and on acquiring an educational goal for 40 Veterans with PTSD who are randomly assigned to an intervention group (N=20) that receives a weekly supported education intervention and a control group that receives services as usual plus an hour of attentive intervention not focused on education.

Aim 2. To examine whether the supported education intervention has secondary effects for improving PTSD symptoms and attitudes on recovery. Objective: Conduct pre- and post assessments of recovery attitudes and of PTSD symptoms, and then compare the control and intervention group for changes in these scores.

Aim 3. To acquire additional process information on the design and implementation of a supported education service necessary for a successful larger trial. Objective: Conduct a process evaluation of the implementation strategies for: participant recruitment, participant drop-out, technician training procedures, technician recovery promoting competence, and curriculum content and pacing using a standardized assessment, exit interviews, peer notes and study records.

ELIGIBILITY:
Inclusion Criteria:

* PTSD
* OIF/OEF Service

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marsha Langer Ellison, PhD MSW, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

REFERENCES:
- [Result] Ellison ML, Mueller L, Smelson D, Corrigan PW, Torres Stone RA, Bokhour BG, Najavits LM, Vessella JM, Drebing C. Supporting the education goals of post-9/11 veterans with self-reported PTSD symptoms: a needs assessment. Psychiatr Rehabil J. 2012 Winter;35(3):209-17. doi: 10.2975/35.3.2012.209.217. PMID 22246119

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans were referred to the study by clinicians and other sources such as Veterans Upward Program and were consented and baselined over a 9 month period.
Groups:
- General Peer Support: Veterans received peer services that did not address educational goals
Period: Overall Study
Arm/Group | Supported Education | General Peer Support
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Supported Education: Rehabilitation counseling using peers to achieve educational goals
- Active Control: Veterans recived peer services that did not address educational goals
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Active Control | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Full Range); unit: years] | 29 [23 to 37] | 29 [21 to 36] | 29 [21 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 15 | 15 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 12 | 14 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: "Supported Education Process Measure"
Description: Number of quarter hours spent in activities related to acquiring an education goal e.g., preparing applications, attending classes. Hours will be logged on a tally sheet adapted from the "Supported Education Process Measure" (Corrigan, 2009).
Time Frame: 6 months
Population: Comparison of means
Measure: Mean (Standard Deviation); unit: number of quarter hours
Groups:
- Supported Education: Supported Education: Rehabilitation counseling using peers to achieve educational goals Intervention group
- General Peer Support: Matched peer attention no supported education service
Arm/Group | Supported Education | General Peer Support
Number analyzed (Participants) | 17 | 16
number of quarter hours | 26.2 (50.2) | 8.2 (21.5)
Statistical Analysis 1: Comparison: Supported Education; Test type: Superiority or Other; p = 0.0059, t-test, 2 sided; Mean Difference (Net) = 18.0, 95% CI 2-sided [14 to 38], Standard Deviation 33.9

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Active Control: Veterans received matched peer attention that did not address educational goals
Arm/Group | Arm 1 | Active Control
Serious Adverse Events (participants affected / at risk) | 2/17 | 0/16
Other Adverse Events (participants affected / at risk) | 7/17 | 3/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=17) | Active Control (N=16)
hospitalization (Psychiatric disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=17) | Active Control (N=16)
discharged from domiciliary (Psychiatric disorders) | 3 (3) | 3 (3)
incarceration (Psychiatric disorders) | 1 (1) | 0 (0)
higher level of care (Psychiatric disorders) | 2 (2) | 0 (0)
back injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes